CLINICAL TRIAL: NCT06535737
Title: A Phase 2, Single Arm Study of Cabozantinib in Patients With Hepatocellular Carcinoma Who Have Received Prior Atezolizumab and Bevacizumab
Acronym: CPAB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: onco-059/67
Record Dates: First submitted 2024-07-24; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; Cabozantinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cabozantinib (Experimental): Open-labelled
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib (Cabometyx) 60, 40 and 20 mg

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common liver cancer and a leading cancer death worldwide. Currently, atezolizumab and bevacizumab combination is the standard of care for patients with advanced HCC. There have not been proven therapy for patients with advanced HCC previously treated with atezolizumab and bevacizumab. Cabozantinib is a proven therapy for patients with advanced HCC previously treated with sorafenib. The study aims to demonstrate the efficacy and safety of cabozantinib in patients with advanced previously treated with atezolziumab and bevacizumab. It is a multi-center single-arm study which all participants will receive cabozantinib. Participants will continue cabozantinib until. disease progression or unacceptable toxicities.

DETAILED DESCRIPTION:
Currently, atezolizumab and bevacizumab combination is the standard of care for patients with advanced HCC. There have not been proven therapy for patients with advanced HCC previously treated with atezolizumab and bevacizumab. Cabozantinib is a proven therapy for patients with advanced HCC previously treated with sorafenib. The study aims to demonstrate the efficacy and safety of cabozantinib in patients with advanced previously treated with atezolziumab and bevacizumab.

This is a phase II, single-arm, multi-center trial which all participants will receive cabozantinib. Eligible patients will provide informed consent to participate the trial. The study will enroll 40 patients. All participants will receive cabozantinib until disease progression or unacceptable toxicities. Efficacy assessment will be performed with CT scan or MRI every 8 weeks. Clinical assessments and laboratory tests will be scheduled every 2-4 weeks for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Radiological, histological or cytological diagnosis of HCC
* The subject has disease that is not amenable to a curative treatment approach (eg, transplant, surgery, radiofrequency ablation)
* Received prior atezolizumab and bevacizumab
* Progression following atezolizumab and bevacizumab treatment for advanced HCC
* Recovery to ≤ Grade 1 from toxicities related to any prior treatments, unless the adverse events are clinically nonsignificant and/or stable on supportive therapy
* Age ≥ 18 years old on the day of consent
* ECOG performance status of 0 or 1
* Adequate hematologic function, based upon meeting the following laboratory criteria within 7 days before enrollment:

  * absolute neutrophil count (ANC) ≥ 1200/mm3 (≥ 1.2 x 109/L)
  * platelets ≥ 60,000/mm3 (≥ 60 x 109/L)
  * hemoglobin ≥ 8 g/dL (≥ 80 g/L)
* Adequate renal function, based upon meeting the following laboratory criteria within 7 days before enrollment:

  * serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockroft-Gault equation: (140 - age) x weight (kg)/(serum creatinine × 72 [mg/dL]) for males. (For females multiply by 0.85.) AND
  * urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1g
* Child-Pugh Score of A or B7
* Total bilirubin ≤ 2 mg/dL (≤ 34.2 μmol/L) within 7 days before enrollment
* Serum albumin ≥ 2 g/dL (≥ 20 g/L) within 7 days before enrollment
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5.0 upper limit of normal (ULN) within 7 days before enrollment
* Hemoglobin A1c (HbA1c) ≤ 8% within 7 days before enrollment
* Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
* Capable of understanding and complying with the protocol requirements and signed informed consent
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression, low body weight, or other reasons.

Exclusion Criteria:

* • Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
* Receipt of more than one prior systemic therapy for advanced HCC. Additional prior systemic therapies used as adjuvant or local therapy are allowed.
* Any type of anticancer agent (including investigational) within 2 weeks before enrollment
* Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment (eg, I-131 or Y-90) within 6 weeks of enrollment. Subject is excluded if there are any clinically relevant ongoing complications from prior radiation therapy.
* Prior cabozantinib treatment
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before enrollment. Eligible subjects must be without corticosteroid treatment at the time of enrollment.
* Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel). Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low-dose LMWH are permitted.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including
  * Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias
* Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment
* Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months before enrollment
* Thromboembolic event within 3 months before enrollment. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible

  o Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
* Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
* Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before enrollment, Note: Complete healing of an intra-abdominal abscess must be confirmed prior to enrollment

  * Major surgery within 2 months before enrollment. Complete healing from major surgery must have occurred 1 month before enrollment. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before enrollment. Subjects with clinically relevant complications from prior surgery are not eligible
  * Cavitating pulmonary lesion(s) or endobronchial disease
  * Lesion invading a major blood vessel (eg, pulmonary artery or aorta)
  * Clinically significant bleeding risk including the following within 3 months of enrollment: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
  * Other clinically significant disorders such as:
* Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)-related illness
* Serious non-healing wound/ulcer/bone fracture
* Malabsorption syndrome
* Uncompensated/symptomatic hypothyroidism
* Requirement for hemodialysis or peritoneal dialysis
* History of solid organ transplantation
* 9. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding are excluded with the following clarification: subjects with history of prior variceal bleeding must have been treated with adequate endoscopic therapy without any evidence of recurrent bleeding for at least 6 months prior to study entry and must be stable on optimal medical management (e.g. non-selective beta blocker, proton pump inhibitor) at study entry.
* Moderate or severe ascites
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 7 days before enrollment
* Note: If the QTcF is > 500 ms in first ECG, a total of 3 ECGs should be performed. If the average of these 3 consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
* Inability to swallow tablets
* Previously identified allergy or hypersensitivity to components of the study treatment formulations
* Pregnant or lactating females
* Diagnosis of another malignancy within 2 years before enrollment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) per RECIST 1.1 at 4th month | 4th month of treatment
  Proportion of participants with stable disease, partial response and complete response at 4th month of cabozantinib treatment based on RECIST 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST 1.1 at 4th month | 4th month of treatment
  Proportion of participants with partial response or complete response at 4th month of treatment based on RECIST 1.1
Progression-free survival (PFS) per RECIST 1.1 | Time from treatment initiation to documented disease progression per RECIST 1.1 or death, whichever came first, assessed up to 24 months
  Time from treatment initiation to documented disease progression per RECIST 1.1 or death
Overall survival (OS) | Time from treatment initiation to patient death, assessed up to 36 months
  Time from treatment initiation to patient death

CONTACTS AND LOCATIONS:
Overall Officials: Suebpong Tanasanvimon, M.D., Study Chair — Chulalongkorn University; Nuttapong Ngamphaiboon, M.D., Principal Investigator — Marisol University; Krittaya Korphaisarn, M.D., Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Abou-Alfa GK, Meyer T, Cheng AL, El-Khoueiry AB, Rimassa L, Ryoo BY, Cicin I, Merle P, Chen Y, Park JW, Blanc JF, Bolondi L, Klumpen HJ, Chan SL, Zagonel V, Pressiani T, Ryu MH, Venook AP, Hessel C, Borgman-Hagey AE, Schwab G, Kelley RK. Cabozantinib in Patients with Advanced and Progressing Hepatocellular Carcinoma. N Engl J Med. 2018 Jul 5;379(1):54-63. doi: 10.1056/NEJMoa1717002. PMID 29972759
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Kelley RK, Rimassa L, Cheng AL, Kaseb A, Qin S, Zhu AX, Chan SL, Melkadze T, Sukeepaisarnjaroen W, Breder V, Verset G, Gane E, Borbath I, Rangel JDG, Ryoo BY, Makharadze T, Merle P, Benzaghou F, Banerjee K, Hazra S, Fawcett J, Yau T. Cabozantinib plus atezolizumab versus sorafenib for advanced hepatocellular carcinoma (COSMIC-312): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Aug;23(8):995-1008. doi: 10.1016/S1470-2045(22)00326-6. Epub 2022 Jul 4. PMID 35798016
- [Background] Rumgay H, Arnold M, Ferlay J, Lesi O, Cabasag CJ, Vignat J, Laversanne M, McGlynn KA, Soerjomataram I. Global burden of primary liver cancer in 2020 and predictions to 2040. J Hepatol. 2022 Dec;77(6):1598-1606. doi: 10.1016/j.jhep.2022.08.021. Epub 2022 Oct 5. PMID 36208844
- [Background] Gherardi E, Birchmeier W, Birchmeier C, Vande Woude G. Targeting MET in cancer: rationale and progress. Nat Rev Cancer. 2012 Jan 24;12(2):89-103. doi: 10.1038/nrc3205. PMID 22270953
- [Background] Kaposi-Novak P, Lee JS, Gomez-Quiroz L, Coulouarn C, Factor VM, Thorgeirsson SS. Met-regulated expression signature defines a subset of human hepatocellular carcinomas with poor prognosis and aggressive phenotype. J Clin Invest. 2006 Jun;116(6):1582-95. doi: 10.1172/JCI27236. Epub 2006 May 18. PMID 16710476
- [Background] You H, Ding W, Dang H, Jiang Y, Rountree CB. c-Met represents a potential therapeutic target for personalized treatment in hepatocellular carcinoma. Hepatology. 2011 Sep 2;54(3):879-89. doi: 10.1002/hep.24450. Epub 2011 Jul 19. PMID 21618573
- [Background] Santoro A, Rimassa L, Borbath I, Daniele B, Salvagni S, Van Laethem JL, Van Vlierberghe H, Trojan J, Kolligs FT, Weiss A, Miles S, Gasbarrini A, Lencioni M, Cicalese L, Sherman M, Gridelli C, Buggisch P, Gerken G, Schmid RM, Boni C, Personeni N, Hassoun Z, Abbadessa G, Schwartz B, Von Roemeling R, Lamar ME, Chen Y, Porta C. Tivantinib for second-line treatment of advanced hepatocellular carcinoma: a randomised, placebo-controlled phase 2 study. Lancet Oncol. 2013 Jan;14(1):55-63. doi: 10.1016/S1470-2045(12)70490-4. Epub 2012 Nov 20. PMID 23182627
- [Background] Greten TF, Korangy F, Manns MP, Malek NP. Molecular therapy for the treatment of hepatocellular carcinoma. Br J Cancer. 2009 Jan 13;100(1):19-23. doi: 10.1038/sj.bjc.6604784. Epub 2008 Nov 18. PMID 19018262
- [Background] You WK, Sennino B, Williamson CW, Falcon B, Hashizume H, Yao LC, Aftab DT, McDonald DM. VEGF and c-Met blockade amplify angiogenesis inhibition in pancreatic islet cancer. Cancer Res. 2011 Jul 15;71(14):4758-68. doi: 10.1158/0008-5472.CAN-10-2527. Epub 2011 May 25. PMID 21613405
- [Background] Sennino B, Ishiguro-Oonuma T, Wei Y, Naylor RM, Williamson CW, Bhagwandin V, Tabruyn SP, You WK, Chapman HA, Christensen JG, Aftab DT, McDonald DM. Suppression of tumor invasion and metastasis by concurrent inhibition of c-Met and VEGF signaling in pancreatic neuroendocrine tumors. Cancer Discov. 2012 Mar;2(3):270-87. doi: 10.1158/2159-8290.CD-11-0240. Epub 2012 Feb 24. PMID 22585997
- [Background] Yakes FM, Chen J, Tan J, Yamaguchi K, Shi Y, Yu P, Qian F, Chu F, Bentzien F, Cancilla B, Orf J, You A, Laird AD, Engst S, Lee L, Lesch J, Chou YC, Joly AH. Cabozantinib (XL184), a novel MET and VEGFR2 inhibitor, simultaneously suppresses metastasis, angiogenesis, and tumor growth. Mol Cancer Ther. 2011 Dec;10(12):2298-308. doi: 10.1158/1535-7163.MCT-11-0264. Epub 2011 Sep 16. PMID 21926191